CLINICAL TRIAL: NCT04430322
Title: Coronavirus Disease 2019 (Covid-19) at the Regional Hospital Center Metz-Thionville: a Descriptive Study
Brief Title: Covid-19 at the Regional Medical Center Metz-Thionville: a Descriptive Study
Acronym: COMETE-19
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02Obs-CHRMT
Record Dates: First submitted 2020-06-11; First posted 2020-06-12 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2022-08

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
France and especially the region "Grand Est" have been damaged by the COVID-19 pandemic. This pandemic resulted in a reorganization of the hospitalization sectors.

In order to better understand the disease, the investigators wish to carry out a descriptive analysis of hospitalized patient data. This study would notably allow us to identify some prognostic factors.

The main objective of this study is to identify individual factors that are associated with a poor prognosis (with ICU admission or death).

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in COVID Unit at the Regional Hospital Center Metz-Thionville during the COVID 19 pandemic
* PCR positive or COVID confirmed with clinical evidence and CT scan

Exclusion Criteria:

* Patients not willing to participate via using their medical files
* Patient transferred after a brief stay in another hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient hospitalized in COVID Unit at the Regional Hospital Center Metz-Thionville during the COVID-19 pandemic with a PCR positive or COVID confirmed with clinical evidence and CT scan.
Sampling Method: Non-Probability Sample
Enrollment: 1045 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
ICU admission | Day 1
  Number of ICU admission during the hospitalization

SECONDARY OUTCOMES:
Hospitalization | Day 1
  The duration of the hospitalization
Length of stay at the ICU | Day 1
  The duration of stay at the ICU
Death | Day 1
  The occurrence of death during the stay
CT scan result | Day 1
  Evocative CT scan result
C reactive protein | Day 1
  C reactive protein value
Blood Count | Day 1
  Blood Count value
Sodium | Day 1
  Sodium value
Urea | Day 1
  Urea value
Troponine | Day 1
  Troponine value via biological data
Liver function | Day 1
  Transaminases value
Coagulation test | Day 1
  Quick test result
Creatinine | day 1
  creatinine value
Clearance | day 1
  creatinine clearance value
Potassium | day 1
  potassium value
Calcium | day 1
  calcium value
Gamma-glutamyl transpeptidase | day 1
  Gamma-glutamyl transpeptidase value
Bilirubine | day 1
  Bilirubine value
Alcaline phosphatase | Day 1
  Alcaline phosphatase value
Prothrombine | Day 1
  Prothrombine value

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Metz Thionville, Metz, France

REFERENCES:
- [Derived] Louis G, Dinot V, Belveyre T, Dirand O, Dunand P, Cadoz C, Gaci R, Gette S, Perez P, Goetz C, Picard Y, Mellati N. Comparison of fully-vaccinated and non/partially-vaccinated critically-ill COVID-19 patients in terms of disease severity: a retrospective observational study. BMC Infect Dis. 2025 Oct 31;25(1):1457. doi: 10.1186/s12879-025-11904-4. PMID 41174545